CLINICAL TRIAL: NCT02192957
Title: Developing a Standardized Atrial Fibrillation Cardioversion Protocol
Brief Title: The Ottawa AF Cardioversion Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: David Birnie (Other)
Responsible Party: Sponsor-Investigator, David Birnie, BSc (Hons), MB ChB, MRCP(UK), MD, Ottawa Heart Institute Research Corporation
Organization: Ottawa Heart Institute Research Corporation (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20140415; Form ID 2788 (Other: Ottawa Health Science Network Research Ethics Board)
Record Dates: First submitted 2014-07-11; First posted 2014-07-17 (Estimated); Last update posted 2019-10-02 (Actual); Status verified 2019-09

CONDITIONS: Atrial Fibrillation
Keywords: cardioversion; electrical cardioversion; atrial fibrillation; cardioversion protocol
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ottawa AF Cardioversion (Other): elective electrical cardioversion for atrial fibrillation (AF) using the Ottawa AF protocol
  Interventions: Device: Lifepak 20E Defibrillator, Licence No: 61944

INTERVENTIONS:
Device: Lifepak 20E Defibrillator, Licence No: 61944 — Intervention will be carried out using Health Canada approved devices for electrical cardioversion, following the steps pre-specified in the Ottawa AF Protocol.
  Ottawa AF Cardioversion
  Other Names: -HEARTSTART XL, Licence No: 24413.; -Kendall 1010P Multi-function Defibrillation Electrodes, Licence No: 21857

SUMMARY:
Atrial fibrillation is an abnormal heart rhythm in which the top chambers of the heart (the atrial chambers) beat very fast. Electrical cardioversion is a technique to convert heart rhythm from AF to normal rhythm. The technique sends out a brief electric shock to the heart through electrodes (paddles or skin patches) applied to the outside of the chest wall. The shock resets the heart rhythm back to its normal pattern.

This technique is practiced at many hospitals, including the Heart Institute, and is not experimental. However no detailed national or international guidelines exist to assist physicians in performing cardioversion. Physicians use a variety of methods. Electrical cardioversion does not always restore normal rhythm. Adjusting the electrical energy dose, changing the electrode position and applying pressure to the electrodes may improve the success rate.

This study will look at the safety and efficacy of a protocol (step by step method) for electrical cardioversion. The protocol prescribes the electrical energy dose, the electrode position and the application of pressure to the electrodes the physician will use. The individual elements of the protocol (energy dose, electrode position and pressure application) are often used by physician in clinical practice but not necessarily in the step by step order.

The purpose of this study is to get all doctors to follow a standard protocol 'the Ottawa AF cardioversion protocol'. We think that using this protocol will improve overall cardioversion success rates. The results of this study may change usual practice in Canada and in other countries.

All supplies, equipment and medications used in the protocol cardioversion are approved by Health Canada.

We estimate that 389 participants from the University of Ottawa Heart Institute will be enrolled in the study over the next 2 years. The results will be compared with a group of previous patients.

DETAILED DESCRIPTION:
Study design:

All eligible and consenting patients will undergo elective electrical cardioversion for atrial fibrillation (AF) using the Ottawa AF protocol.The fact that the physician follows the protocol makes this experimental. Aside from following the protocol, subjects will receive standard care before, during and after the procedure. Outcomes of the procedure and clinical features know to affect cardioversion efficacy will be collected. These will be compared to a group of 500 previous patients who underwent elective electrical cardioversion for AF at the Heart Institute.

Methodology:

The Ottawa AF protocol prescribes the electrical energy dose, the electrode position and the application of pressure to the electrodes the physician will use. The individual elements of the protocol (energy dose, electrode position and pressure application) are often used by physician in clinical practice but not necessarily in the step by step order.

The Ottawa AF protocol prescribes the following:

* the starting energy dose (200 J) and electrode placement (anterior-posterior)
* the second electrode placement (anterior-lateral) if the first shock is not successful
* addition of pressure to electrodes if second shock is not successful
* step up of energy dose (360 J) along with pressure to electrodes if third shock is not successful
* optional further steps at physician's choice if fourth shock is not successful

ELIGIBILITY:
Inclusion Criteria:

* Documented atrial fibrillation within last 12 months
* On continuous systemic oral anticoagulation for 28 days prior to the day of cardioversion or must have undergone a recent (< 48 hrs) trans-esophageal echocardiogram prior to the day of cardioversion
* Able to provide informed consent

Exclusion Criteria:

* Presence of intracardiac thrombus
* Pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 389 (Actual)
Dates: Start 2015-08; Primary Completion 2017-12 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Last shock efficacy | immediately after cardioversion
  Last shock efficacy defined as success ( two or more beats of sinus rhythm) or failure.

OTHER OUTCOMES:
Adverse Events | participants will be followed for the duration of hospital stay for elective cardioversion, an expected average of 2 hours.
  adverse events related to cardioversion

CONTACTS AND LOCATIONS:
Overall Officials: David H Birnie, MD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- University of Ottawa Heart Institution, Ottawa, Ontario, Canada

REFERENCES:
- [Result] Ramirez FD, Sadek MM, Boileau I, Cleland M, Nery PB, Nair GM, Redpath CJ, Green MS, Davis DR, Charron K, Henne J, Zakutney T, Beanlands RSB, Hibbert B, Wells GA, Birnie DH. Evaluation of a novel cardioversion intervention for atrial fibrillation: the Ottawa AF cardioversion protocol. Europace. 2019 May 1;21(5):708-715. doi: 10.1093/europace/euy285. PMID 30535367